CLINICAL TRIAL: NCT04365153
Title: Canakinumab to Reduce Deterioration of Cardiac and Respiratory Function in SARSCoV2 Associated Acute Myocardial Injury With Heightened Inflammation
Brief Title: Canakinumab in Covid-19 Cardiac Injury (The Three C Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IND 149328
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Results first posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: COVID-19; SARS-CoV 2
MeSH Terms: conditions — COVID-19 | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High Dose Intervention (Active Comparator): 600 mg of canakinumab (8 mg/kg for patients </= 40 kg)
  Interventions: Drug: Canakinumab Injection 600mg
- Low Dose Intervention (Active Comparator): 300 mg of canakinumab (4 mg/kg for patients </= 40 kg)
  Interventions: Drug: Canakinumab Injection 300mg
- Control (Placebo Comparator): Placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Canakinumab Injection 600mg — Subjects will be given one-time intravenous infusion of 600 mg of canakinumab (8 mg/kg for patients </= 40 kg) in 250 mL of 5% dextrose infused IV over 2 hours
  Other Names: ACZ885
  Arms: High Dose Intervention
Drug: Canakinumab Injection 300mg — Subjects will be given one-time intravenous infusion of 300 mg of canakinumab (4 mg/kg for patients </= 40 kg) in 250 mL of 5% dextrose infused IV over 2 hours
  Other Names: ACZ885
  Arms: Low Dose Intervention
Drug: Placebos — 250 mL of 5% dextrose infused IV over 2 hours
  Other Names: Control
  Arms: Control

SUMMARY:
TThe purpose of this prospective, Phase 2, single center, blinded, randomized controlled study is to demonstrate as a proof of concept that early treatment with canakinumab prevents progressive heart and respiratory failure in patients with COVID-19 infection. These results will lead to and inform a Phase III randomized placebo-controlled trial.

DETAILED DESCRIPTION:
This is a prospective, Phase 2, single center, blinded randomized-controlled study designed as a proof of concept to demonstrate that early treatment with canakinumab prevents progressive heart and respiratory failure in patients with COVID 19 infection, myocardial injury and hyperinflammation. These results will lead to a Phase III randomized placebo-controlled trial.

The study will be performed in approximately 7 months total, starting from the first patient enrolled with enrollment expected to complete within 2 months. The follow-up period is 5 months for each patient enrolled. The end of the study, including statistical analysis and drafting of the final report is expected within 1 month from the last patient enrolled.

A total of 45 patients will be randomized using a 1:1:1 allocation ratio: 15 subjects will receive 600 mg intravenous canakinumab (8 mg/kg if </= 40 kg), 15 subjects will receive 300 mg intravenous canakinumab (4 mg/kg if </= 40 kg), and 15 patients will receive placebo infusion.

The investigator, clinical team, and subject will be blinded to treatment assignment.

ELIGIBILITY:
Inclusion Criteria: Subjects eligible for inclusion in this study must meet all of the following criteria:

1. Written informed consent must be obtained before any assessment is performed
2. Hospitalized due to COVID-19 infection
3. Documented SARS-CoV2 acute myocardial injury: Defined as upper respiratory tract specimen positive for COVID-19 AND Troponin T greater than 99th percentile upper reference range without signs or symptoms of acute myocardial ischemia
4. NT-proBNP greater than the age-adjusted upper reference limit
5. Receiving current standard therapy
6. C-reactive protein (CRP) > 50 mg/L

Exclusion Criteria: Subjects meeting any of the following criteria are not eligible for inclusion in this study.

1. Alternative explanation for acute cardiac injury (Type I or Type II MI according to 4th Universal Definition of Myocardial Infarction, which in addition to a rise and fall of troponin above the 99th percentile upper reference limit, includes symptoms of acute myocardial ischemia, new ischemic ECG changes, development of pathologic Q waves, and imaging evidence of damage in a pattern consistent with an ischemic etiology)
2. Chronic Systolic Heart Failure with EF<35%
3. Age < 18 years-old
4. Uncontrolled systemic bacterial or fungal infection
5. Concomitant viral infection (e.g., Influenza or other respiratory virus)
6. Pregnant. Breast-feeding women are eligible with the decision to continue or discontinue breast-feeding during therapy taking into account the risk of infant exposure, the benefits of breast-feeding to the infant, and benefits of treatment to the mother.
7. On mechanical circulatory support
8. On mechanical ventilation for greater than 48 hours
9. Resuscitated cardiac arrest
10. Has a known hypersensitivity to canakinumab or any of its excipients
11. Neutrophil count <1000/mm3
12. Has a history of myeloproliferative disorder or active malignancy receiving chemotherapy
13. Known active tuberculosis or history of incompletely treated tuberculosis
14. Current treatment with immunosuppressive agents
15. Chronic prednisone use >10 mg/daily (for more than 3 weeks prior to admission)
16. Has a history of solid-organ or bone marrow transplant
17. Severe pre-existing liver disease with clinically significant portal hypertension
18. End-stage renal disease on chronic renal replacement therapy
19. Enrollment in another investigational study using immunosuppressive therapy
20. In the opinion of the investigator and clinical team, should not participate in the study
21. If male and sexually active, must have documented vasectomy or must practice birth control and not donate sperm during the study and for 3 months after study drug administration.
22. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of investigational drug. Such methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject
    * Use of oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul C Cremer, M. D., Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cleveland Clinic Florida, Weston, Florida
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Dose Intervention | Low Dose Intervention | Control
Started | 15 | 14 | 16
Completed | 15 | 14 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Intervention | Low Dose Intervention | Control | Total
Number analyzed (Participants) | 15 | 14 | 16 | 45
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66.4 [63.5 to 72.9] | 70.7 [64.7 to 74.6] | 68.2 [56.1 to 83.3] | 68.8 [61.1 to 74.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 3 | 12
  Male | 11 | 9 | 13 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 8 | 4 | 5 | 17
  Caucasian | 6 | 9 | 10 | 25
  Asian | 0 | 1 | 0 | 1
  Hispanic | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 16 | 45
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 29.2 [28.0 to 46.4] | 28.3 [25.8 to 32.0] | 29.2 [24.0 to 42.9] | 28.8 [25.3 to 36.3]
Diabetes mellitus [Count of Participants; unit: Participants] | 10 | 4 | 7 | 21
Hypertension [Count of Participants; unit: Participants] | 11 | 9 | 12 | 32
Hyperlipidemia [Count of Participants; unit: Participants] | 12 | 8 | 9 | 29
Coronary Artery Disease [Count of Participants; unit: Participants] | 2 | 4 | 4 | 10
Stroke [Count of Participants; unit: Participants] | 0 | 1 | 1 | 2
Atrial fibrillation or flutter [Count of Participants; unit: Participants] | 2 | 2 | 2 | 6
COPD [Count of Participants; unit: Participants] | 3 | 3 | 2 | 8
Chronic kidney disease [Count of Participants; unit: Participants] | 6 | 2 | 7 | 15
Current or former smoker [Count of Participants; unit: Participants] | 5 | 4 | 6 | 15
Time from symptoms onset to randomization [Median (Inter-Quartile Range); unit: days] | 6 [3 to 8] | 9 [6 to 11] | 6 [4 to 10] | 7 [4 to 9]
Dyspnea [Count of Participants; unit: Participants] | 11 | 11 | 14 | 36
Temperature [Median (Inter-Quartile Range); unit: degrees Celsius] | 36.8 [36.6 to 37.2] | 37.4 [36.9 to 37.9] | 36.8 [36.5 to 36.9] | 36.9 [36.6 to 37.4]
Hospitalized requiring invasive mechanical ventilation [Count of Participants; unit: Participants] | 5 | 2 | 3 | 10
Hospitalized requiring nasal high-flow oxygen or non-invasive ventilation, or both [Count of Participants; unit: Participants] | 3 | 3 | 5 | 11
Hospitalized requiring supplemental oxygen [Count of Participants; unit: Participants] | 5 | 9 | 6 | 20
Hospitalized, not requiring supplemental oxygen [Count of Participants; unit: Participants] | 2 | 0 | 2 | 4
Baseline PaO2/FiO2 ratio [Median (Inter-Quartile Range); unit: ratio] | 148 [73 to 203] | 160 [77 to 246] | 117 [66 to 210] | 148 [73 to 204]
Baseline SOFA scores (SOFA: Sequential organ failure assessment) [Median (Inter-Quartile Range); unit: score on a scale] — SOFA score is the Sequential Organ Failure Assessment which measures dysfunction within PaO2/FIO2 Factor, Platelets Factor, Total Bilirubin Factor, Blood Pressure, Glasgow Coma Score Factor and Renal Factor, each on a scale of 0 (normal function) to 4 (severe dysfunction). The total minimum score is 0, the total maximum score is 24, with higher scores indicating severe dysfunction.
  score on a scale | 3 [2 to 6] | 2 [2 to 4] | 4 [2 to 5] | 3 [2 to 5]
Corticosteroids [Count of Participants; unit: Participants] | 8 | 3 | 10 | 21
Remdesivir [Count of Participants; unit: Participants] | 10 | 5 | 6 | 21
High sensitivity troponin T (ng/L) (reference range <12 ng/L) [Median (Inter-Quartile Range); unit: ng/L] | 21 [15 to 31] | 25 [14 to 36] | 32 [16 to 163] | 22 [15 to 37]
N-terminal pro B-type natriuretic peptide (pg/mL) (reference range <125 pg/mL) [Median (Inter-Quartile Range); unit: pg/mL] | 371 [181 to 1401] | 372 [277 to 1508] | 810 [349 to 10264] | 479 [248 to 1508]
C reactive protein (mg/dL) (reference range 0.0-0.4 mg/dL) [Median (Inter-Quartile Range); unit: mg/dL] | 12.7 [10.8 to 19.7] | 12.2 [6.4 to 15.3] | 17.6 [15.0 to 19.9] | 15.3 [12.1 to 18.5]
Lymphocyte count (reference range 1.0-4.0 k/uL) [Median (Inter-Quartile Range); unit: k/uL] | 0.8 [0.7 to 1.0] | 0.7 [0.5 to 1.2] | 0.5 [0.4 to 0.9] | 0.7 [0.5 to 1.0]
Ferritin (ng/mL)(reference range 14.7-205.1 ng/mL) [Median (Inter-Quartile Range); unit: ng/mL] | 740 [448 to 1969] | 998 [857 to 1626] | 1246 [768 to 2355] | 1015 [589 to 2111]
D-dimer (ng/mL)(reference range <500 ng/mL) [Median (Inter-Quartile Range); unit: ng/mL] | 1795 [870 to 3430] | 950 [730 to 1340] | 1500 [560 to 3340] | 1320 [730 to 2140]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Improvement at Day 14
Description: Number of patients with either an improvement of two points on a seven category ordinal scale or discharge from the hospital
Time Frame: Up to day 14
Measure: Count of Participants; unit: Participants
Groups:
- Control: Placebo: 250 mL of 5% dextrose infused IV over 2 hours
Arm/Group | High Dose Intervention | Low Dose Intervention | Control
Number analyzed (Participants) | 15 | 14 | 16
Participants | 9 | 7 | 9

2. Secondary Outcome: All-cause Mortality
Description: Number of patients who expired after treatment
Time Frame: Up to day 28
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Intervention | Low Dose Intervention | Control
Number analyzed (Participants) | 15 | 14 | 16
Participants | 1 | 3 | 3

ADVERSE EVENTS:
Time Frame: 150 days
Arm/Group | High Dose Intervention | Low Dose Intervention | Control
All-Cause Mortality (participants affected / at risk) | 1/15 | 3/14 | 4/16
Serious Adverse Events (participants affected / at risk) | 5/15 | 6/14 | 7/16
Other Adverse Events (participants affected / at risk) | 11/15 | 11/14 | 11/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Intervention (N=15) | Low Dose Intervention (N=14) | Control (N=16)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (3)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Liver Dysfunction (Hepatobiliary disorders) | 0 (0) | 1 (2) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Shock (General disorders) | 1 (1) | 3 (4) | 1 (1)
Superinfection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clot (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Breakdown (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased Platelet Count (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Fungemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertensive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ventilator Tube Occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0)
DVT (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Intervention (N=15) | Low Dose Intervention (N=14) | Control (N=16)
Acute Kidney Injury (Renal and urinary disorders) | 4 (4) | 5 (5) | 6 (9)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 4 (7)
Arrhythmia (Cardiac disorders) | 2 (2) | 2 (3) | 2 (2)
Bleeding (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1)
Encephalitis/Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Liver Dysfunction (Hepatobiliary disorders) | 0 (0) | 4 (4) | 5 (5)
Pneumonia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Shock (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hypophosphatemia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Clot (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Elevated Ferritin (Investigations) | 2 (2) | 5 (5) | 5 (5)
Hypotension (Cardiac disorders) | 1 (1) | 2 (2) | 4 (4)
Elevated CRP (Investigations) | 2 (2) | 6 (6) | 3 (3)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (General disorders) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hypovolemia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rigors (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Restless Leg Syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathic Lower Extremity Pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
UTI (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)
Positive Respiratory Culture (Infections and infestations) | 2 (2) | 0 (0) | 2 (4)
Skin Breakdown (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Worsening D-Dimer (Investigations) | 2 (2) | 5 (5) | 3 (3)
Fever (General disorders) | 2 (2) | 3 (3) | 4 (4)
Corneal Abrasion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
COVID 19 Hyperinflammation (Infections and infestations) | 0 (0) | 1 (2) | 3 (3)
Elevated ANC (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Elevated WBC (Investigations) | 0 (0) | 0 (0) | 2 (2)
Elevated LD (Investigations) | 0 (0) | 2 (2) | 3 (3)
Worsening of Hemoglobin and Hematocrit (Investigations) | 1 (1) | 2 (3) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Stidor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flash Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Elevated Cardiac Enzymes (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT04365153/Prot_SAP_000.pdf